CLINICAL TRIAL: NCT05122065
Title: Defining the Vaginal Microbiome and the Vaginal pH of Menopausal Women With and Without Genitourinary Syndrome and With and Without Hormone Replacement Therapy
Brief Title: Menopausal Vaginal Microbiome
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: FemTec Health Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: MENO0721
Record Dates: First submitted 2021-11-04; First posted 2021-11-16 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Menopause; Hormone Replacement Therapy; Genitourinary Syndrome of Menopause
Keywords: vaginal microbiome; menopause; hormone replacement therapy; Genitourinary syndrome of menopause

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Asymptomatic/non-HRT: Samples derived from women in menopause who do not self-reportedly experience GSM (Genitourinary Syndrome of Menopause) and who do not take HRT (Hormone Replacement Therapy).
- Asymptomatic/HRT: Samples derived from women in menopause who do not self-reportedly experience GSM and who take HRT
- GSM/non-HRT: Samples derived from women in menopause who self-reportedly experience GSM and who do not take HRT
- GSM/HRT: Samples derived from women in menopause who self-reportedly experience GSM and who take HRT

SUMMARY:
In this study the investigators will analyze the vaginal microbiome of menopausal women in order to shed light on its potential implication on menopausal symptoms and quality of life. Moreover, the investigators will assess the effect of hormone replacement treatment on symptoms and overall quality of life during menopause and whether women under hormone replacement treatment have distinct vaginal microbiome profiles.

ELIGIBILITY:
Inclusion Criteria:

* Women who are females from birth
* Women between 40-70 years old
* Women that are US residents, understand, and speak English
* Women of all race and ethnicities
* Women that are postmenopausal (at least 12 consecutive months without a period)
* Women with a naturally occuring menopause
* Women willing to abstain from all sexual activity, feminine hygiene products (eg. douches, wipes, washes, sprays, powders, moisturizers/lubricants, deodorant suppositories, tablet suppositories, anti-itch creams, hot tubs) on the vaginal area, and any vaginal suppositories for 48 hours before sampling
* Women who are healthy (without GSM)
* Women who have GSM:

  1. with formal diagnosis of GSM, or
  2. who regularly experience a couple of the following symptoms: (i) vaginal dryness, vaginal burning, vaginal discharge & genital itching, vaginal irritation, (ii) light bleeding, discomfort or pain during or after intercourse, decreased lubrication during intercourse, decreased arousal, orgasm, libido, (iii) painful or difficult urination (dysuria), urinary frequency and urgency, recurrent UTIs (Urinary Tract Infections).
* Women who either take or do not take HRT, including estrogen-only medicines, combination of estrogen/progestin medicines, combination of estrogen/other medicines.

Exclusion Criteria:

* Women suffering from gynecological diseases including polycystic ovary syndrome, endometriosis, pelvic inflammatory disease, active HPV (human papillomavirus) or herpes simplex virus in the past few months, BV (Bacterial Vaginosis), yeast infections, or positive for any STD (Sexually Transmitted Disease; genital warts, chlamydia, gonorrhea, syphilis, trichomoniasis), HIV (Human Immunodeficiency Virus), cancer, type I diabetes, type II diabetes, chronic kidney disease.
* Women having any genital surgery including removal of one or both ovaries, uterus or cervix.
* Women whose menopause occurred by surgical operation (hysterectomy, oophorectomy), or drug/treatment (eg. chemotherapy, radiation therapy).
* Women using douches daily or weekly.
* Women who use on a regular basis one of the following: metformin, antihistamines, antidepressants, corticosteroids, boric acid, laxatives, antifungal/antimycotic medication.
* Women using any oral or vaginal prebiotics, probiotics, or antibiotics in the past 6 months.
* Women who take progestin-only medicines including progestin-only HRT.

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women who are females from birth
Study Population: Participants will be postmenopausal women with or without self-reported GSM that either follow or do not follow an HRT plan.
Sampling Method: Non-Probability Sample
Enrollment: 432 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-12-15 (Estimated)

PRIMARY OUTCOMES:
Vaginal microbiome sample collection | Baseline
  Identify microbiome-based bacterial signatures to distinguish the different menopausal groups and the CST (Community State Type) group clustering according to the vaginal microbiome of menopausal women.

SECONDARY OUTCOMES:
Demographic questionnaire | Baseline
  Data will include ethnic/cultural background, body weight, and height, age, sexual orientation, relationship status, education status/academic background, employment status, current occupation, area of residence, chronic condition(s), number of children, and type of birth given, age of last period, last Pap test and thyroid test, contraception method, use of prescription or non-prescription medications and supplements, smoking and alcohol habits, dietary habits, information source about menopause, attitude towards talking about menopause, self-image and changes on hair/skin/nails, dental health and body weight during menopause, awareness of menopause state, online services/app or products used during menopause, delivery address for testing kits.
Day-to-Day Impact of Vaginal Aging (DIVA) questionnaire | Baseline
  Participants will answer a questionnaire including four multi-item scales addressing symptoms impact on: 1) activities of daily living, 2) emotional well-being, 3) sexual functioning, and 4) self-concept and body image. The possible score range for all domain scales is 0 to 4, with higher scores denoting greater impact of vaginal symptoms.
Menopause Rating Scale (MRS) questionnaire | Baseline
  Participants will answer the 11-question questionnaire regarding the presence or absence and intensity of their menopause-related symptoms. The minimum value is zero and the maximum is four with the latter indicating very severe symptoms.
Brief Resilience Scale (BRS) questionnaire | Baseline
  Participants will answer a 6-question questionnaire concerning their ability to recover from stress. This questionnaire has two types of questions namely, one with positive meaning in which the scoring scale is from 1 (strongly disagree) to 5 (strongly agree) and the second one has negative meaning with the scoring scale ranging from 1 (strongly agree) to 5 (strongly disagree).
Vaginal pH -at home test kit | Baseline
  Participants will be asked to take a vaginal pH sample in duplicate. Participants will be asked to fill in a form with their vaginal pH test results obtained from the vaginal pH test.
Facial Skin Type Test | Baseline
  The facial skin type testing kit (USP Solutions, Klagenfurt, Austria) will include two "Skin Oil Tester Sebutapes", a skin test results template, and a product insert with useful information and instructions for the participants.
Body Hydration Test | Baseline
  Participants will be asked to take the body hydration test once on their hand and once on their leg. The body hydration testing kit (USP Solutions, Klagenfurt, Austria) will include two "Dry Skin Test D-Squames", a skin test results template, and a product insert with useful information and instructions for the participants.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Capone, PhD, Principal Investigator — FemTec Health Inc.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Farage MA, Miller KW, Sobel JD. Dynamics of the vaginal ecosystem - hormonal influences. Infectious Diseases: Research and Treatment. 2010. doi: 10.4137/IDRT.S3903
- [Background] Gliniewicz K, Schneider GM, Ridenhour BJ, Williams CJ, Song Y, Farage MA, Miller K, Forney LJ. Comparison of the Vaginal Microbiomes of Premenopausal and Postmenopausal Women. Front Microbiol. 2019 Feb 14;10:193. doi: 10.3389/fmicb.2019.00193. eCollection 2019. PMID 30837959
- [Background] Muhleisen AL, Herbst-Kralovetz MM. Menopause and the vaginal microbiome. Maturitas. 2016 Sep;91:42-50. doi: 10.1016/j.maturitas.2016.05.015. Epub 2016 Jun 1. PMID 27451320
- [Background] Angelou K, Grigoriadis T, Diakosavvas M, Zacharakis D, Athanasiou S. The Genitourinary Syndrome of Menopause: An Overview of the Recent Data. Cureus. 2020 Apr 8;12(4):e7586. doi: 10.7759/cureus.7586. PMID 32399320
- [Background] Lobo RA. Hormone-replacement therapy: current thinking. Nat Rev Endocrinol. 2017 Apr;13(4):220-231. doi: 10.1038/nrendo.2016.164. Epub 2016 Oct 7. PMID 27716751
- [Background] Nguyen TM, Do TTT, Tran TN, Kim JH. Exercise and Quality of Life in Women with Menopausal Symptoms: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Int J Environ Res Public Health. 2020 Sep 26;17(19):7049. doi: 10.3390/ijerph17197049. PMID 32993147
- [Background] Gloor GB, Macklaim JM, Pawlowsky-Glahn V, Egozcue JJ. Microbiome Datasets Are Compositional: And This Is Not Optional. Front Microbiol. 2017 Nov 15;8:2224. doi: 10.3389/fmicb.2017.02224. eCollection 2017. PMID 29187837
- [Background] Hillmann B, Al-Ghalith GA, Shields-Cutler RR, Zhu Q, Gohl DM, Beckman KB, Knight R, Knights D. Evaluating the Information Content of Shallow Shotgun Metagenomics. mSystems. 2018 Nov 13;3(6):e00069-18. doi: 10.1128/mSystems.00069-18. eCollection 2018 Nov-Dec. PMID 30443602
- [Background] Yang Q, Wang Y, Wei X, Zhu J, Wang X, Xie X, Lu W. The Alterations of Vaginal Microbiome in HPV16 Infection as Identified by Shotgun Metagenomic Sequencing. Front Cell Infect Microbiol. 2020 Jun 23;10:286. doi: 10.3389/fcimb.2020.00286. eCollection 2020. PMID 32656096
- [Background] Oliver A, LaMere B, Weihe C, Wandro S, Lindsay KL, Wadhwa PD, Mills DA, Pride DT, Fiehn O, Northen T, de Raad M, Li H, Martiny JBH, Lynch S, Whiteson K. Cervicovaginal Microbiome Composition Is Associated with Metabolic Profiles in Healthy Pregnancy. mBio. 2020 Aug 25;11(4):e01851-20. doi: 10.1128/mBio.01851-20. PMID 32843557
- [Background] Feehily C, Crosby D, Walsh CJ, Lawton EM, Higgins S, McAuliffe FM, Cotter PD. Shotgun sequencing of the vaginal microbiome reveals both a species and functional potential signature of preterm birth. NPJ Biofilms Microbiomes. 2020 Nov 12;6(1):50. doi: 10.1038/s41522-020-00162-8. PMID 33184260
- [Background] Nappi RE, Martini E, Cucinella L, Martella S, Tiranini L, Inzoli A, Brambilla E, Bosoni D, Cassani C, Gardella B. Addressing Vulvovaginal Atrophy (VVA)/Genitourinary Syndrome of Menopause (GSM) for Healthy Aging in Women. Front Endocrinol (Lausanne). 2019 Aug 21;10:561. doi: 10.3389/fendo.2019.00561. eCollection 2019. PMID 31496993
- [Background] Jenabi E, Shobeiri F, Hazavehei SM, Roshanaei G. Assessment of Questionnaire Measuring Quality of Life in Menopausal Women: A Systematic Review. Oman Med J. 2015 May;30(3):151-6. doi: 10.5001/omj.2015.34. PMID 26171119
- [Background] Davis SR, Lambrinoudaki I, Lumsden M, Mishra GD, Pal L, Rees M, Santoro N, Simoncini T. Menopause. Nat Rev Dis Primers. 2015 Apr 23;1:15004. doi: 10.1038/nrdp.2015.4. PMID 27188659
- [Background] Whiteley J, DiBonaventura Md, Wagner JS, Alvir J, Shah S. The impact of menopausal symptoms on quality of life, productivity, and economic outcomes. J Womens Health (Larchmt). 2013 Nov;22(11):983-90. doi: 10.1089/jwh.2012.3719. Epub 2013 Oct 1. PMID 24083674
- [Background] Portman DJ, Gass ML; Vulvovaginal Atrophy Terminology Consensus Conference Panel. Genitourinary syndrome of menopause: new terminology for vulvovaginal atrophy from the International Society for the Study of Women's Sexual Health and the North American Menopause Society. Menopause. 2014 Oct;21(10):1063-8. doi: 10.1097/GME.0000000000000329. PMID 25160739
- [Background] The NAMS 2020 GSM Position Statement Editorial Panel. The 2020 genitourinary syndrome of menopause position statement of The North American Menopause Society. Menopause. 2020 Sep;27(9):976-992. doi: 10.1097/GME.0000000000001609. PMID 32852449
- [Background] Briggs P. Genitourinary syndrome of menopause. Post Reprod Health. 2020 Jun;26(2):111-114. doi: 10.1177/2053369119884144. Epub 2019 Oct 23. PMID 31645194
- [Background] Castelo-Branco C, Biglia N, Nappi RE, Schwenkhagen A, Palacios S. Characteristics of post-menopausal women with genitourinary syndrome of menopause: Implications for vulvovaginal atrophy diagnosis and treatment selection. Maturitas. 2015 Aug;81(4):462-9. doi: 10.1016/j.maturitas.2015.05.007. Epub 2015 May 30. PMID 26071816
- [Background] Barrientos-Duran A, Fuentes-Lopez A, de Salazar A, Plaza-Diaz J, Garcia F. Reviewing the Composition of Vaginal Microbiota: Inclusion of Nutrition and Probiotic Factors in the Maintenance of Eubiosis. Nutrients. 2020 Feb 6;12(2):419. doi: 10.3390/nu12020419. PMID 32041107
- [Background] Godha K, Tucker KM, Biehl C, Archer DF, Mirkin S. Human vaginal pH and microbiota: an update. Gynecol Endocrinol. 2018 Jun;34(6):451-455. doi: 10.1080/09513590.2017.1407753. Epub 2017 Dec 22. PMID 29271266
- [Background] Kiss H, Kogler B, Petricevic L, Sauerzapf I, Klayraung S, Domig K, Viernstein H, Kneifel W. Vaginal Lactobacillus microbiota of healthy women in the late first trimester of pregnancy. BJOG. 2007 Nov;114(11):1402-7. doi: 10.1111/j.1471-0528.2007.01412.x. Epub 2007 Sep 17. PMID 17877778
- [Background] Juliana NCA, Suiters MJM, Al-Nasiry S, Morre SA, Peters RPH, Ambrosino E. The Association Between Vaginal Microbiota Dysbiosis, Bacterial Vaginosis, and Aerobic Vaginitis, and Adverse Pregnancy Outcomes of Women Living in Sub-Saharan Africa: A Systematic Review. Front Public Health. 2020 Dec 10;8:567885. doi: 10.3389/fpubh.2020.567885. eCollection 2020. PMID 33363078
- [Background] Ceccarani C, Foschi C, Parolin C, D'Antuono A, Gaspari V, Consolandi C, Laghi L, Camboni T, Vitali B, Severgnini M, Marangoni A. Diversity of vaginal microbiome and metabolome during genital infections. Sci Rep. 2019 Oct 1;9(1):14095. doi: 10.1038/s41598-019-50410-x. PMID 31575935
- [Background] Mendling, W. Normal and abnormal vaginal microbiota. LaboratoriumsMedizin. 2016; 40(4): 239-246. doi: 10.1515/labmed-2016-0011
- [Background] Superti F, De Seta F. Warding Off Recurrent Yeast and Bacterial Vaginal Infections: Lactoferrin and Lactobacilli. Microorganisms. 2020 Jan 17;8(1):130. doi: 10.3390/microorganisms8010130. PMID 31963487
- [Background] Amabebe E, Anumba DOC. The Vaginal Microenvironment: The Physiologic Role of Lactobacilli. Front Med (Lausanne). 2018 Jun 13;5:181. doi: 10.3389/fmed.2018.00181. eCollection 2018. PMID 29951482
- [Background] Qi W, Li H, Wang C, Li H, Fan A, Han C, Xue F. The effect of pathophysiological changes in the vaginal milieu on the signs and symptoms of genitourinary syndrome of menopause (GSM). Menopause. 2020 Aug 17;28(1):102-108. doi: 10.1097/GME.0000000000001644. PMID 32810079
- [Background] Brotman RM, Shardell MD, Gajer P, Fadrosh D, Chang K, Silver MI, Viscidi RP, Burke AE, Ravel J, Gravitt PE. Association between the vaginal microbiota, menopause status, and signs of vulvovaginal atrophy. Menopause. 2014 May;21(5):450-8. doi: 10.1097/GME.0b013e3182a4690b. PMID 24080849
- [Background] Shen J, Song N, Williams CJ, Brown CJ, Yan Z, Xu C, Forney LJ. Effects of low dose estrogen therapy on the vaginal microbiomes of women with atrophic vaginitis. Sci Rep. 2016 Apr 22;6:24380. doi: 10.1038/srep24380. PMID 27103314
- [Background] Geng L, Huang W, Jiang S, Zheng Y, Zhou Y, Zhou Y, Hu J, Li P, Tao M. Effect of Menopausal Hormone Therapy on the Vaginal Microbiota and Genitourinary Syndrome of Menopause in Chinese Menopausal Women. Front Microbiol. 2020 Nov 20;11:590877. doi: 10.3389/fmicb.2020.590877. eCollection 2020. PMID 33329470
- [Background] Mitchell CM, Srinivasan S, Zhan X, Wu MC, Reed SD, Guthrie KA, LaCroix AZ, Fiedler T, Munch M, Liu C, Hoffman NG, Blair IA, Newton K, Freeman EW, Joffe H, Cohen L, Fredricks DN. Vaginal microbiota and genitourinary menopausal symptoms: a cross-sectional analysis. Menopause. 2017 Oct;24(10):1160-1166. doi: 10.1097/GME.0000000000000904. PMID 28640154
- [Background] Hummelen R, Macklaim JM, Bisanz JE, Hammond JA, McMillan A, Vongsa R, Koenig D, Gloor GB, Reid G. Vaginal microbiome and epithelial gene array in post-menopausal women with moderate to severe dryness. PLoS One. 2011;6(11):e26602. doi: 10.1371/journal.pone.0026602. Epub 2011 Nov 2. PMID 22073175
- [Background] Ma ZS, Li L. Quantifying the human vaginal community state types (CSTs) with the species specificity index. PeerJ. 2017 Jun 27;5:e3366. doi: 10.7717/peerj.3366. eCollection 2017. PMID 28674641
- [Background] Ginkel PD, Soper DE, Bump RC, Dalton HP. Vaginal flora in postmenopausal women: the effect of estrogen replacement. Infect Dis Obstet Gynecol. 1993;1(2):94-7. doi: 10.1155/S1064744993000225. PMID 18475325
- [Background] Heinemann C, Reid G. Vaginal microbial diversity among postmenopausal women with and without hormone replacement therapy. Can J Microbiol. 2005 Sep;51(9):777-81. doi: 10.1139/w05-070. PMID 16391657
- [Background] Nelson HD. Commonly used types of postmenopausal estrogen for treatment of hot flashes: scientific review. JAMA. 2004 Apr 7;291(13):1610-20. doi: 10.1001/jama.291.13.1610. PMID 15069049
- [Background] Galhardo CL, Soares JM Jr, Simoes RS, Haidar MA, Rodrigues de Lima G, Baracat EC. Estrogen effects on the vaginal pH, flora and cytology in late postmenopause after a long period without hormone therapy. Clin Exp Obstet Gynecol. 2006;33(2):85-9. PMID 16903243
- [Background] Setty P, Rekedal L, Warren MP. Vaginal estrogen use and effects on quality of life and urogenital morbidity in postmenopausal women after publication of the Women's Health Initiative in New York City. Menopause. 2016 Jan;23(1):7-10. doi: 10.1097/GME.0000000000000493. PMID 26263282
- [Background] Quince C, Walker AW, Simpson JT, Loman NJ, Segata N. Shotgun metagenomics, from sampling to analysis. Nat Biotechnol. 2017 Sep 12;35(9):833-844. doi: 10.1038/nbt.3935. PMID 28898207
- [Background] Rausch P, Ruhlemann M, Hermes BM, Doms S, Dagan T, Dierking K, Domin H, Fraune S, von Frieling J, Hentschel U, Heinsen FA, Hoppner M, Jahn MT, Jaspers C, Kissoyan KAB, Langfeldt D, Rehman A, Reusch TBH, Roeder T, Schmitz RA, Schulenburg H, Soluch R, Sommer F, Stukenbrock E, Weiland-Brauer N, Rosenstiel P, Franke A, Bosch T, Baines JF. Comparative analysis of amplicon and metagenomic sequencing methods reveals key features in the evolution of animal metaorganisms. Microbiome. 2019 Sep 14;7(1):133. doi: 10.1186/s40168-019-0743-1. PMID 31521200
- [Background] Durazzi F, Sala C, Castellani G, Manfreda G, Remondini D, De Cesare A. Comparison between 16S rRNA and shotgun sequencing data for the taxonomic characterization of the gut microbiota. Sci Rep. 2021 Feb 4;11(1):3030. doi: 10.1038/s41598-021-82726-y. PMID 33542369
- [Background] Ravel J, Gajer P, Abdo Z, Schneider GM, Koenig SS, McCulle SL, Karlebach S, Gorle R, Russell J, Tacket CO, Brotman RM, Davis CC, Ault K, Peralta L, Forney LJ. Vaginal microbiome of reproductive-age women. Proc Natl Acad Sci U S A. 2011 Mar 15;108 Suppl 1(Suppl 1):4680-7. doi: 10.1073/pnas.1002611107. Epub 2010 Jun 3. PMID 20534435
- [Background] Mancabelli L, Tarracchini C, Milani C, Lugli GA, Fontana F, Turroni F, van Sinderen D, Ventura M. Vaginotypes of the human vaginal microbiome. Environ Microbiol. 2021 Mar;23(3):1780-1792. doi: 10.1111/1462-2920.15441. Epub 2021 Feb 28. PMID 33615652
- [Background] Beck D, Foster JA. Machine learning techniques accurately classify microbial communities by bacterial vaginosis characteristics. PLoS One. 2014 Feb 3;9(2):e87830. doi: 10.1371/journal.pone.0087830. eCollection 2014. PMID 24498380
- [Background] Pérez-Gómez JF, Canul-Reich J, Hernández-Torruco J, Hernández-Ocaña B. Predictor selection for bacterial vaginosis diagnosis using decision tree and relief algorithms. Applied Sciences. 2020; 10(9):3291. doi: 10.3390/app10093291
- [Background] Lee YH, Kang GU, Jeon SY, Tagele SB, Pham HQ, Kim MS, Ahmad S, Jung DR, Park YJ, Han HS, Shin JH, Chong GO. Vaginal Microbiome-Based Bacterial Signatures for Predicting the Severity of Cervical Intraepithelial Neoplasia. Diagnostics (Basel). 2020 Nov 26;10(12):1013. doi: 10.3390/diagnostics10121013. PMID 33256024
- [Background] Loomba R, Seguritan V, Li W, Long T, Klitgord N, Bhatt A, Dulai PS, Caussy C, Bettencourt R, Highlander SK, Jones MB, Sirlin CB, Schnabl B, Brinkac L, Schork N, Chen CH, Brenner DA, Biggs W, Yooseph S, Venter JC, Nelson KE. Gut Microbiome-Based Metagenomic Signature for Non-invasive Detection of Advanced Fibrosis in Human Nonalcoholic Fatty Liver Disease. Cell Metab. 2019 Sep 3;30(3):607. doi: 10.1016/j.cmet.2019.08.002. No abstract available. PMID 31484056
- [Background] Li J, Zhao F, Wang Y, Chen J, Tao J, Tian G, Wu S, Liu W, Cui Q, Geng B, Zhang W, Weldon R, Auguste K, Yang L, Liu X, Chen L, Yang X, Zhu B, Cai J. Gut microbiota dysbiosis contributes to the development of hypertension. Microbiome. 2017 Feb 1;5(1):14. doi: 10.1186/s40168-016-0222-x. PMID 28143587
- [Background] Armour CR, Nayfach S, Pollard KS, Sharpton TJ. A Metagenomic Meta-analysis Reveals Functional Signatures of Health and Disease in the Human Gut Microbiome. mSystems. 2019 May 14;4(4):e00332-18. doi: 10.1128/mSystems.00332-18. eCollection 2019 Jul-Aug. PMID 31098399
- [Background] Lloyd-Price J, Mahurkar A, Rahnavard G, Crabtree J, Orvis J, Hall AB, Brady A, Creasy HH, McCracken C, Giglio MG, McDonald D, Franzosa EA, Knight R, White O, Huttenhower C. Strains, functions and dynamics in the expanded Human Microbiome Project. Nature. 2017 Oct 5;550(7674):61-66. doi: 10.1038/nature23889. Epub 2017 Sep 20. PMID 28953883
- [Background] Huang AJ, Gregorich SE, Kuppermann M, Nakagawa S, Van Den Eeden SK, Brown JS, Richter HE, Walter LC, Thom D, Stewart AL. Day-to-Day Impact of Vaginal Aging questionnaire: a multidimensional measure of the impact of vaginal symptoms on functioning and well-being in postmenopausal women. Menopause. 2015 Feb;22(2):144-54. doi: 10.1097/GME.0000000000000281. PMID 24983271
- [Background] Heinemann LA, Potthoff P, Schneider HP. International versions of the Menopause Rating Scale (MRS). Health Qual Life Outcomes. 2003 Jul 30;1:28. doi: 10.1186/1477-7525-1-28. PMID 12914663
- [Background] Smith BW, Dalen J, Wiggins K, Tooley E, Christopher P, Bernard J. The brief resilience scale: assessing the ability to bounce back. Int J Behav Med. 2008;15(3):194-200. doi: 10.1080/10705500802222972. PMID 18696313
- [Background] Tsementzi D, Pena-Gonzalez A, Bai J, Hu YJ, Patel P, Shelton J, Dolan M, Arluck J, Khanna N, Conrad L, Scott I, Eng TY, Konstantinidis KT, Bruner DW. Comparison of vaginal microbiota in gynecologic cancer patients pre- and post-radiation therapy and healthy women. Cancer Med. 2020 Jun;9(11):3714-3724. doi: 10.1002/cam4.3027. Epub 2020 Apr 1. PMID 32237205
- [Background] Lee JE, Lee S, Lee H, Song YM, Lee K, Han MJ, Sung J, Ko G. Association of the vaginal microbiota with human papillomavirus infection in a Korean twin cohort. PLoS One. 2013 May 22;8(5):e63514. doi: 10.1371/journal.pone.0063514. Print 2013. PMID 23717441
- [Background] Wang X, Ji X. Sample Size Estimation in Clinical Research: From Randomized Controlled Trials to Observational Studies. Chest. 2020 Jul;158(1S):S12-S20. doi: 10.1016/j.chest.2020.03.010. PMID 32658647